CLINICAL TRIAL: NCT03974737
Title: Evaluation of the Compensatory Reserve Index and Psychosocial Factors in Pediatric Autonomic Dysfunction
Brief Title: CRI in POTS in Adolescents
Acronym: POTS
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 18-2618
Record Dates: First submitted 2019-05-24; First posted 2019-06-05 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: POTS; Postural Orthostatic Tachycardia Syndrome; Dysautonomia; CRI; Compensatory Reserve Index
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Autonomic Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Adolescents with POTS: Adolescents with Postural Orthostatic Tachycardia Syndrome (POTS) who meet diagnostic criteria for an orthostatic heart rate increase of >30, between ages 12-21 are eligible for this group. They will have a urine specific gravity conducted at the beginning of the clinic visit to assess hydration status. If urine specific gravity shows adequate hydration, subjects will proceed with orthostatic measurements with concomitant CRI measurements (via a non-invasive pulse oximetry monitor). (Subjects who are dehydrated will be given electrolyte drinks for rehydration and urine specific gravity will be rechecked after survey completion and before CRI and orthostatic measurements.) Following the CRI and orthostatic measurements, subjects and their parents will be asked to complete a series of surveys via REDcap.
  Interventions performed:
  * Urine specific gravity measurement
  * CRI measurements, orthostatic vitals measurements
  * Survey administration
  Interventions: Device: CRI device (non-invasive vitals sign measurement)
- Adolescents without POTS, Control Group: Adolescents without Postural Orthostatic Tachycardia Syndrome (POTS) between ages 12-21 are eligible for this group. This group of subjects will have a urine specific gravity conducted at the beginning of the clinic visit to assess hydration status. If the urine specific gravity shows adequate hydration, subjects will proceed with orthostatic measurements with concomitant CRI measurements (via a non-invasive pulse oximetry monitor). (Subjects who are dehydrated will be given electrolyte drinks for rehydration and their urine specific gravity will be rechecked after survey completion and before CRI and orthostatic measurements.) Following the CRI and orthostatic measurements, subjects and their parents will be asked to complete a series of surveys via REDcap.
  Interventions performed:
  * Urine specific gravity measurement
  * CRI measurements, orthostatic vitals measurements
  * Survey administration
  Interventions: Device: CRI device (non-invasive vitals sign measurement)
- Adolescents diagnosed with POTS who do not meet HR: Adolescents diagnosed with Postural Orthostatic Tachycardia Syndrome (POTS) between ages 12-21, who do not meet diagnostic heart rate criteria, are eligible for this group. This group of subjects will have a urine specific gravity conducted at beginning of the clinic visit to assess hydration status. If the urine specific gravity shows adequate hydration, subjects will proceed with orthostatic measurements with concomitant CRI measurements (via a non-invasive pulse oximetry monitor). (Subjects who are dehydrated will be given electrolyte drinks for rehydration and urine specific gravity will be rechecked after survey completion and before CRI and orthostatic measurements.) Following the CRI and orthostatic measurements, subjects and their parents will be asked to complete a series of surveys via REDcap.
  Interventions performed:
  * Urine specific gravity measurement
  * CRI measurements, orthostatic vitals measurements
  * Survey administration
  Interventions: Device: CRI device (non-invasive vitals sign measurement)

INTERVENTIONS:
Device: CRI device (non-invasive vitals sign measurement) — Survey administration, Orthostatic vital measurements
  Other Names: Survey administration, Orthostatic vital measurements

SUMMARY:
The investigators aim to study whether the Compensatory Reserve Index (CRI) (an FDA approved device that assesses intravascular volume) can be used to evaluate severity of Postural Orthostatic Tachycardia Syndrome (POTS) and whether the CRI value has a correlation with severity of psychosocial symptoms and functional impairment associated with POTS.

DETAILED DESCRIPTION:
Autonomic dysfunction (or dysautonomia) describes several medical conditions linked to the autonomic nervous system. One of these is Postural Orthostatic Tachycardia Syndrome (POTS). In pediatric populations, symptoms of autonomic dysfunction include an increase in heart rate when standing up (tachycardia), dizziness, nausea, vomiting, fatigue, headaches, abdominal discomfort, and sleep disturbances. POTS is specifically characterized by orthostatic intolerance and a forty beats per minute (bpm) increase in heart rate upon standing. The etiology of POTS is poorly understood, and there is limited literature on the management of POTS in pediatric populations. In the U.S., POTS is estimated to affect 1-3 million people.

The ability of the CRI algorithm to accurately distinguish individuals with varying tolerances to reduced central blood volume can be attributed to a unique function of the algorithm, which analyzes and compares the entirety of each waveform in a window of time to trend subtle features that correspond with varying degrees of central volume loss. CRI can also detect vascular changes associated with postural orthostatic tachycardia syndrome. CRI will be evaluated in subjects at supine and standing positions along with traditional orthostatic measures.

Following CRI measurements, subjects and their parents will be asked to complete a series of surveys to assess their psychosocial symptoms and functional impairment. The CRI measurement and survey completion will occur over the course of one clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent participants must be aged 12 to 21 years (inclusive).
* Each participant must have at one parent/legal guardian who can provide informed consent for the adolescent and participate in the study by completing study questionnaires.
* Moreover, as the majority of study measures are only validated for use in English, only English-speaking patients will be included in this study.

Exclusion Criteria:

* Adolescents will be excluded from the study if they are outside the age range of 12-21 years old
* Adolescents who are wards of the state
* Adolescents who are incarcerated
* Adolescents who are decisionally impaired (i.e., have difficulty understanding the protocol during the consent process, and/or research team member is unsure of individual's ability to correctly identify whether the research study would need to stop or not)
* Adolescents who object at any time to participating in the study
* Adolescents who have a pacemaker
* Adolescents who are taking beta blocker medications
* Adolescents who were were hospitalized in the past month for serious medical conditions affecting their cardiopulmonary system (note, this does not include recent hospitalizations for trauma or burns).
* Adolescents will also be excluded if their parent/legal guardian(s) are unwilling to participate in the study and/or do not have legal custody of the adolescent participant.
* Adolescents who do not speak English will be excluded from the study as majority of the study measures are only validated in English.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will include adolescents with POTS 12-21 years old and adolescents without POTS 12-21 years old. One parent will be required to attend the study visit.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Change in Compensatory Reserve Index (CRI) Values | Minute 1 through minute 20
  This is a value between 0 and 1. The CRI values will be noted from minute 1 to minute 20. This study has only one visit.
Physical Symptoms Score as assessed by a Survey | 1 day (study visit)
  Subjects will complete a survey to assess severity of physical symptoms (fatigue, dizziness, weakness, headache, chest pain, palpitations, sweating, shortness of breath, abdominal pain, nausea, vomiting, period pain, cries easily, altered temperature, discoloration of extremities, peripheral edema, numbness, brain fog, diarrhea, constipation, blurred vision, muscle pain, joint pain, exercise intolerance, insomnia, joint hypermobility, sensitivity to light, early society, etc.). Possible scores range from 0 to 10, with 10 indicating the most severe/debilitating symptoms and 0 indicating no physical symptoms/normal functionality. The survey will be completed during the study visit. This study has only one visit.
Frequency of Anxiety in Days as assessed by a Survey | 1 day (study visit)
  Subjects will complete a survey to assess how frequently (how many days) they experienced feelings of acute anxiety over the past month. The survey will be completed during the study visit. This study has only one visit.
Hypermobility as evaluated by the Beighton scale | 1 day (study visit)
  The Beighton Score is a validated measure used to evaluate hypermobility in children on a scale of 0-9 for different joints using 3 score bands. A higher Beighton score is associated with hypermobility. The assessment will be completed during the study visit. This study has only one visit.
Frequency of Feelings of Stress in Days as assessed by a survey | 1 day (study visit)
  Subjects will complete a survey to assess how frequently (how many days) they experienced feelings of stress over the past month. The survey will be completed during the study visit. This study has only one visit.
Frequency of difficulty with sleep as assessed by a survey | 1 day (study visit)
  Subjects will complete a survey to assess how long it takes them to fall asleep, how often they wake up, how long it takes to fall back asleep after waking up, and the frequency of difficulties with sleep.The survey will be completed during the study visit. This study has only one visit.
Revised Child Anxiety and Depression Scale (RCADS and RCADS-P) | 1 day (study visit)
  Subjects and their parent(s) will complete this well-established survey tool to assess the frequency of symptoms of anxiety and depression. The survey will be completed during the study visit. This study has only one visit.
Functional disability inventory (FDI) | 1 day (study visit)
  Participants and their parent(s) will be asked to complete a 15-question survey to evaluate the difficulty of daily tasks with a scale of impossible (4), a lot of trouble (3), some trouble (2), a little trouble (1), and no trouble (0) (39). This measure will be adapted very slightly to reflect the ubiquity of electronic media for today's adolescents, i.e., question 11 will be modified from "Watching TV" to "Watching TV and other screens." This measure yields an overall summed score. The survey will be completed during the study visit. This study has only one visit.
Social Connectedness Scale | 1 day (study visit)
  The Social Connectedness Scale, developed by Lee, assesses the responder's perceptions of social connectedness (i.e., the perception of interpersonal closeness with the social world) through 15 self-report items. The assessment will be completed during the study visit. This study has only one visit.
Friendship scale | 1 day (study visit)
  The "Close Friend Support/Regard" subscale of the Social Support Scale for Children and Adolescents will be used to assess the adolescent's perception that he/she has a close friend who he/she can tell problems to, who truly understands him/her, who he/she can complain to about things that bother them, who he/she can spend time with, and who really listens to what he/she says. This subscale comprises 6 items rated on a Likert scale from "really true for me" and "sort of true for me" for the positive phrasing of the item (e.g., "Some teenagers have a close friend who really understands them") to "sort of true for me" and "really true for me" for the negative phrasing of the item (e.g., "Other teenagers don't have a close friend who really understands them."). Given that some participants will be above 18 years, we will modify the wording to "some people". The assessment will be completed during the study visit. This study has only one visit.
Frequency of friendship contact | 1 day (study visit)
  Participants will be asked to indicate, over the past month, on how many occasions they have spent time with a close friend outside of school (i.e., free entry). The survey will be completed during the study visit. This study has only one visit.
Family Assessment Device General Functioning scale (GFS) | 1 day (study visit)
  The Family Assessment GFS is a twelve-point scale that evaluates the "overall health or pathology in family functioning" via analysis of six dimensions of family functioning: problem solving, communication, roles, affective responsiveness, affective involvement, and behavior control. This will be completed by subjects and their parent(s). The survey will be completed during the study visit. This study has only one visit.
Sexual maturity Rating (Tanner stage) | 1 day (study visit)
  This questionnaire with image demonstrations of the different Tanner stages will ask patients to self-report their appropriate Tanner stages.The questionnaire will be completed during the study visit. This study has only one visit.
Parent Behavior Adult Responses to Children's Symptoms (ARCS) | 1 day (study visit)
  The ARCS is a 29-point scale with a goal of assessment of parent responses to their children's symptoms (i.e. protectiveness, minimization, encouragement, and monitoring).The assessment will be completed during the study visit. This study has only one visit.
Parent Mental Health- PHQ-9 | 1 day (study visit)
  The Parent Mental Health scales, Parent Health Questionnaire 9 item scale (PHQ-9) and Generalized Anxiety Disorder 7 item scale (GAD-7), are short self-reported questionnaires that are widely used with established psychometrics in the parent population. The PHQ-9 assessment will be completed during the study visit. This study has only one visit.
Parent Mental Health- GAD-7 | 1 day (study visit)
  The Parent Mental Health scales, Parent Health Questionnaire 9 item scale (PHQ-9) and Generalized Anxiety Disorder 7 item scale (GAD-7), are short self-reported questionnaires that are widely used with established psychometrics in the parent population. The GAD-7 assessment will be completed during the study visit. This study has only one visit.

CONTACTS AND LOCATIONS:
Overall Officials: Clio Pitula, PhD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grigoriou E, Boris JR, Dormans JP. Postural orthostatic tachycardia syndrome (POTS): association with Ehlers-Danlos syndrome and orthopaedic considerations. Clin Orthop Relat Res. 2015 Feb;473(2):722-8. doi: 10.1007/s11999-014-3898-x. Epub 2014 Aug 26. PMID 25156902
- [Background] Johnson JN, Mack KJ, Kuntz NL, Brands CK, Porter CJ, Fischer PR. Postural orthostatic tachycardia syndrome: a clinical review. Pediatr Neurol. 2010 Feb;42(2):77-85. doi: 10.1016/j.pediatrneurol.2009.07.002. PMID 20117742
- [Background] Kizilbash SJ, Ahrens SP, Bruce BK, Chelimsky G, Driscoll SW, Harbeck-Weber C, Lloyd RM, Mack KJ, Nelson DE, Ninis N, Pianosi PT, Stewart JM, Weiss KE, Fischer PR. Adolescent fatigue, POTS, and recovery: a guide for clinicians. Curr Probl Pediatr Adolesc Health Care. 2014 May-Jun;44(5):108-33. doi: 10.1016/j.cppeds.2013.12.014. PMID 24819031
- [Background] Boris JR, Bernadzikowski T. Demographics of a large paediatric Postural Orthostatic Tachycardia Syndrome Program. Cardiol Young. 2018 May;28(5):668-674. doi: 10.1017/S1047951117002888. Epub 2018 Jan 23. PMID 29357955
- [Background] Kritzberger CJ, Antiel RM, Wallace DP, Zacharias JD, Brands CK, Fischer PR, Harbeck-Weber C. Functional disability in adolescents with orthostatic intolerance and chronic pain. J Child Neurol. 2011 May;26(5):593-8. doi: 10.1177/0883073810390366. Epub 2011 Feb 7. PMID 21303761
- [Background] Pederson CL, Brook JB. Health-related quality of life and suicide risk in postural tachycardia syndrome. Clin Auton Res. 2017 Apr;27(2):75-81. doi: 10.1007/s10286-017-0399-5. Epub 2017 Feb 6. PMID 28168561
- [Background] Bruce BK, Weiss KE, Harrison TE, Allman DA, Petersen MA, Luedkte CA, Fischer PR. Interdisciplinary Treatment of Maladaptive Behaviors Associated with Postural Orthostatic Tachycardia Syndrome (POTS): A Case Report. J Clin Psychol Med Settings. 2016 Jun;23(2):147-59. doi: 10.1007/s10880-015-9438-3. PMID 26538160
- [Background] Lewis I, Pairman J, Spickett G, Newton JL. Clinical characteristics of a novel subgroup of chronic fatigue syndrome patients with postural orthostatic tachycardia syndrome. J Intern Med. 2013 May;273(5):501-10. doi: 10.1111/joim.12022. Epub 2013 Jan 7. PMID 23206180
- [Background] Convertino VA, Moulton SL, Grudic GZ, Rickards CA, Hinojosa-Laborde C, Gerhardt RT, Blackbourne LH, Ryan KL. Use of advanced machine-learning techniques for noninvasive monitoring of hemorrhage. J Trauma. 2011 Jul;71(1 Suppl):S25-32. doi: 10.1097/TA.0b013e3182211601. PMID 21795890
- [Background] Moulton SL, Mulligan J, Grudic GZ, Convertino VA. Running on empty? The compensatory reserve index. J Trauma Acute Care Surg. 2013 Dec;75(6):1053-9. doi: 10.1097/TA.0b013e3182aa811a. PMID 24256681

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT03974737/Prot_SAP_000.pdf